CLINICAL TRIAL: NCT04960436
Title: Clinical Effect of Allogeneic Meniscus Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200506M
Record Dates: First submitted 2021-06-27; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-06

CONDITIONS: Meniscus Lesion
MeSH Terms: interventions — Meniscectomy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meniscus Allograft Transplantation (Experimental): The patient underwent Meniscus Allograft Transplantation
  Interventions: Procedure: Meniscus Allograft Transplantation
- Meniscectomy (Active Comparator): The patient underwent Meniscectomy
  Interventions: Procedure: Meniscectomy

INTERVENTIONS:
Procedure: Meniscus Allograft Transplantation — patients received surgery of Meniscus Allograft Transplantation
  Arms: Meniscus Allograft Transplantation
Procedure: Meniscectomy — patients received surgery of Meniscectomy
  Arms: Meniscectomy

SUMMARY:
In this study, patients who underwent allogeneic meniscus transplantation and meniscus resection were followed up for more than 10years to evaluate the long-term efficacy and explore the cartilage protective role of meniscus transplantation.

DETAILED DESCRIPTION:
To investigate the long-term clinical effect of allogeneic meniscus transplantation, IKDC score, Lysholom score, Tegner score, VAS score, etc. were used to compare the clinical effects of allogeneic meniscus transplantation, and the progress of knee joint degeneration and cartilage injury was evaluated through X-ray and MRI.

ELIGIBILITY:
Inclusion Criteria:

The age is less than 50 years; the force line is basically normal (≤ ± 3°); the joint is stable or the joint stability is corrected at the same time during the operation; the joint degeneration or large area cartilage damage. In the transplantation group, 10 patients experienced pain or swelling in the joint space of the affected side for an average of 35 months after meniscus resection, and then received meniscus transplantation. The other 8 patients underwent meniscus transplantation at the same time as meniscus resection. Patients in the resection group received meniscus transplantation at the same time. Symptoms, signs, and magnetic resonance imaging (MRI) were diagnosed as a meniscus tear and the judgment during the operation could not be preserved, so a total meniscus was performed.

Exclusion Criteria:

Severe knee synovial disease; severe joint degeneration or extensive cartilage damage; improper force lines; severely unstable joints that cannot be corrected; both meniscuses are removed; the other knee joint has a history of severe trauma or surgery.

Ages: 16 Years to 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2005-02-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Magnetic resonance imaging (MRI) | Before the operation
  All MRI scans were obtained with a 3.0-T MRI scanner (Magnetom Trio with TIM system, Siemens Healthcare). Five routine MRI sequences with a section thickness of 4 mm were obtained in all patients. Preoperative and postoperative evaluations of the articular cartilage of the transplanted compartment were performed with the Yulish score41 (grade 0 = normal; grade 1 = normal contour 6 abnormal signal; grade 2 = superficial fraying, erosion, or ulceration of <50%; grade 3 = partial-thickness defect of >50% but <100%; grade 4 = full-thickness cartilage loss). The signal of the meniscus allograft in the coronal plane of the T2-weighted fast spin echo sequence was graded on a scale of 0 to 3.
Radiographs | 10 years after the operation
  All patients also obtained 45° flexion weightbearing AP radiographs of both the ipsilateral and contralateral sides at final follow-up. The radiograph of the total length of the lower limbs was used to evaluate alignment. In the AP plain radiographs, the shortest distance between the femoral condyle and tibial plateau of the transplanted side was measured and designated as the joint space height. The difference between the ipsilateral and contralateral sides was calculated to identify joint space narrowing. In addition, Kellgren-Lawrence (K-L) grading was used to assess the osteoarthritic status of the knee.
Magnetic resonance imaging (MRI) | 10 years after the operation
  All MRI scans were obtained with a 3.0-T MRI scanner (Magnetom Trio with TIM system, Siemens Healthcare). Five routine MRI sequences with a section thickness of 4 mm were obtained in all patients. Preoperative and postoperative evaluations of the articular cartilage of the transplanted compartment were performed with the Yulish score41 (grade 0 = normal; grade 1 = normal contour 6 abnormal signal; grade 2 = superficial fraying, erosion, or ulceration of <50%; grade 3 = partial-thickness defect of >50% but <100%; grade 4 = full-thickness cartilage loss). The signal of the meniscus allograft in the coronal plane of the T2-weighted fast spin echo sequence was graded on a scale of 0 to 3.
Radiographs | Before the operation
  All patients also obtained 45° flexion weightbearing AP radiographs of both the ipsilateral and contralateral sides at final follow-up. The radiograph of the total length of the lower limbs was used to evaluate alignment. In the AP plain radiographs, the shortest distance between the femoral condyle and tibial plateau of the transplanted side was measured and designated as the joint space height. The difference between the ipsilateral and contralateral sides was calculated to identify joint space narrowing. In addition, Kellgren-Lawrence (K-L) grading was used to assess the osteoarthritic status of the knee.

SECONDARY OUTCOMES:
visual analog scale (VAS) scores | Before and 10 to 15 years after the operation
  visual analog scale (VAS) scores was applied to evaluate knee pain. 0 points means no pain, 10 points means severe pain.
International Knee Documentation Committee (IKDC) score | Before and 10 to 15 years after the operation
  At present, it is recognized internationally that IKDC has relatively high reliability, effectiveness and sensitivity for the assessment of At present, it is recognized internationally that IKDC has relatively high reliability, effectiveness and sensitivity for the assessment of the subjective and objective symptoms of the knee joint system.
Tegner score | Before and 10 to 15 years after the operation
  This score is widely used by exercise assessors for patients with knee joint disease. This scoring method divides the patient's exercise level into 0-10 points, 0 as disability, and 10 as being able to participate in national competitive sports.
Lysholm score | Before and 10 to 15 years after the operation
  This score is often used together with the Tegner score. The scores of this scoring system are generally high and focus more on the assessment of daily activities rather than sports.

CONTACTS AND LOCATIONS:
Overall Officials: Jia-kuo Yu, Prof., Study Chair — Peking University Third Hospital
Locations (1):
- Institute of Sports Medicine, Peking University Third Hospital, Beijing, Beijing Municipality, China